CLINICAL TRIAL: NCT03876158
Title: Transitioning to a Valve -Gated Intrathecal Drug Delivery System (IDDS): An Open-Label, Non-Randomized, Single-Blind, Multi-Center, Cross-Over Study (TRANSIT)
Brief Title: Transitioning to a Valve -Gated Intrathecal Drug Delivery System (IDDS)
Acronym: TRANSIT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study will not be conducted by Dr Lubenow
Sponsor: Rush University Medical Center (Other)
Collaborators: Flowonix Medical (Industry)
Responsible Party: Principal Investigator, Timothy Lubenow, Director, Pain Center, Rush University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ORA# 19011103
Record Dates: First submitted 2019-03-06; First posted 2019-03-15 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain; Intractable Pain; Back Pain
MeSH Terms: conditions — Chronic Pain; Pain, Intractable; Back Pain

STUDY DESIGN:
Intervention Model Description: Prior Peristaltic Synchromed II intrathecal pump's data prior to crossover to valve-gated Flowonix Prometra® II Programmable Pump is recorded to compare.
Who Masked: Participant
Masking Description: This open-label, non-randomized, single-blind, multi-center study is designed to evaluate effects of a planned 20% dose reduction when converting to valve-gated from a peristaltic pump. Study participants will be blinded (single blind) to the dose reduction aspect of this trial and must remain blinded to this dose reduction information throughout the trial in an attempt to provide an unbiased assessment of the pain encountered by the patient with their pain pump medications used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prometra® Programmable Pump (Active Comparator): Pain scores and drug doses will be prospectively collected for valve-gated Prometra® Programmable Pump system(Flowonix Medical)' at (refill #1, refill #2, refill #3) and will be compared to retrospectively collected pain (VAS) scores and drug doses from the last refill prior to peristaltic pump explant.
  Interventions: Device: Prometra II Programmable Pump system(Flowonix Medical)
- Prior records for peristaltic pump (Other): Prior pain scores and drug doses from the patients who need a new valve gated pump will be recorded and used for comparison after it is changed.
  Interventions: Device: Prometra II Programmable Pump system(Flowonix Medical)

INTERVENTIONS:
Device: Prometra II Programmable Pump system(Flowonix Medical) — This valve gated Prometra II Programmable Pump system will be replacing prior peristaltic Synchromed II pump
  Other Names: Prior peristaltic Synchromed II pump

SUMMARY:
Flowonix Prometra® II Programmable Pump may require a smaller dose of drug when converting from other commercially available intrathecal drug delivery systems (IDDS).

DETAILED DESCRIPTION:
This open-label, non-randomized, single-blind, multi-center study is designed to evaluate effects of a planned 20% dose reduction when converting to valve-gated from a peristaltic pump. Study participants will be blinded (single blind) to the dose reduction aspect of this trial and must remain blinded to this dose reduction information throughout the trial in an attempt to provide an unbiased assessment of the pain encountered by the patient with their pain pump medications used.

This study will compare the historical pain medication dose and pain scores using the peristaltic pump at baseline as well as from the last pump refill visit prior to explant to the prospective pain medication dose and pain scores using the valve-gated pump and collected at refill visits 1, 2 and 3 after valve-gated pump implant (but not exceed 12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female between the ages of 22 and 85 years
2. Be capable of giving informed consent and completing assessments required by the study
3. Have pain intensity of greater than 5 out of 10 as measured by VAS
4. Have an active existing peristaltic intrathecal drug delivery system
5. Have stable drug dosage for at least 6 weeks prior to valve-gated pump implant
6. Be an appropriate candidate for surgery
7. Be able to comply with required study visits and assessments including English proficiency

Exclusion Criteria:

1. Have a significant pain disorder not intended to be treated with the test device or comparator
2. Be terminally ill and/or have a life expectancy of less than 6 months
3. Be a pregnant/lactating woman or a woman of child-bearing potential
4. Have a systemic or local infection (contraindicated for pump implantation)
5. Have history/evidence of an active disruptive psychiatric disorder or other known condition with potential to impact compliance with study visits and assessments
6. Have an underlying condition increasing susceptibility to infection

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Reduced pain medication through Prometra Implantable Pump System | 12 months from Implant
  Total consumption of Pain medication both oral and intra thecal would also be recorded to show change in pain medication.

SECONDARY OUTCOMES:
Change in pain score: Visual Analog Scale for Pain | 12 months from Implant
  Visual Analog Scale for Pain is being used assess the pain throughout the 12 month which shows No pain at one end to Pain as bad as it could be at other end.

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Study Chair — Rush University Medical Center; Timothy R Lubenow, MD, Principal Investigator — Rush University Medical Center; Robert McCarthy, D. Pharm, Study Director — Rush University Medical Center
Locations (1):
- Rush University Medical Center Pain Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayek SM, Deer TR, Pope JE, Panchal SJ, Patel VB. Intrathecal therapy for cancer and non-cancer pain. Pain Physician. 2011 May-Jun;14(3):219-48. PMID 21587327
- [Result] Hayek SM, Veizi E, Hanes M. Intrathecal Hydromorphone and Bupivacaine Combination Therapy for Post-Laminectomy Syndrome Optimized with Patient-Activated Bolus Device. Pain Med. 2016 Mar;17(3):561-571. doi: 10.1093/pm/pnv021. Epub 2015 Dec 14. PMID 26814257
- [Result] Konrad PE, Huffman JM, Stearns LM, Plunkett RJ, Grigsby EJ, Stromberg EK, Roediger MP, Wells MD, Weaver TW. Intrathecal Drug Delivery Systems (IDDS): The Implantable Systems Performance Registry (ISPR). Neuromodulation. 2016 Dec;19(8):848-856. doi: 10.1111/ner.12524. Epub 2016 Oct 12. PMID 27730704
- [Result] Tangen KM, Leval R, Mehta AI, Linninger AA. Computational and In Vitro Experimental Investigation of Intrathecal Drug Distribution: Parametric Study of the Effect of Injection Volume, Cerebrospinal Fluid Pulsatility, and Drug Uptake. Anesth Analg. 2017 May;124(5):1686-1696. doi: 10.1213/ANE.0000000000002011. PMID 28431428